CLINICAL TRIAL: NCT07330193
Title: Flowable Resin Composite: In Vitro Investigation of Antibacterial Effect and Calcium & Phosphorus Content and Two-Year Clinical Performance in Class I Restorations
Brief Title: Flowable Resin Composite: Two-Year Clinical Performance in Class I Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: A06080622
Record Dates: First submitted 2025-12-27; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Class I Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- conventional flowable resin composite (Active Comparator)
  Interventions: Procedure: Restoration with CFC
- self adhesive flowable resin composite (Active Comparator)
  Interventions: Procedure: Restoration with SARC
- highly filled flowable resin composite (Active Comparator)
  Interventions: Procedure: Restoration with HFFC
- bioactive self adhesive flowable resin composite (Active Comparator)
  Interventions: Procedure: Restoration with bioactive SARC

INTERVENTIONS:
Procedure: Restoration with CFC — using conventional flowable resin composite materials to restore small occlusal carious lesions
  Arms: conventional flowable resin composite
Procedure: Restoration with HFFC — using highly filled flowable resin composite to restore small class I carious lesions
  Arms: highly filled flowable resin composite
Procedure: Restoration with SARC — using self-adhesive flowable resin composite to restore small class I carious lesions
  Arms: self adhesive flowable resin composite
Procedure: Restoration with bioactive SARC — using bioactive self-adhesive flowable resin composite to restore small class I carious lesions
  Arms: bioactive self adhesive flowable resin composite

SUMMARY:
Evaluating Two-year clinical performance of class I restored with four different flowable resin composite restorations.

ELIGIBILITY:
Inclusion Criteria: •patients with bilateral occlusal small Class I carious lesions

* • Good general health.

  * Patient aging 18-25 year.
  * Patient available for follow-up visits
  * Good oral hygiene

Exclusion Criteria:

Patients with orthodontic treatment

* Severe or chronic periodontitis
* Parafunctional habits
* Sensitivity to resin-based material.
* Poor oral hygiene.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Modified FDI criteria | two years
  successful restorations percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided